CLINICAL TRIAL: NCT02300493
Title: Four Year Weight Change of Cornell Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1108002406
Record Dates: First submitted 2014-11-21; First posted 2014-11-25 (Estimated); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Weight Gain
Keywords: among college students
MeSH Terms: conditions — Weight Gain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental (Experimental): weigh themselves daily
  Interventions: Behavioral: Experimental
- Control (Active Comparator): Weigh themselves every six months
  Interventions: Behavioral: Experimental

INTERVENTIONS:
Behavioral: Experimental — Asked to weigh themselves

SUMMARY:
Examining the effect of daily self-weighing on the ability of student to prevent from gaining weight during their four years at Cornell.

DETAILED DESCRIPTION:
A group of freshman volunteers were randomly assigned to one of two groups. Both groups were given an internet based scale (Withings). The experimental group was asked to weigh themselves daily. The controls were asked to weigh themselves three times within one week every six months in response to being contacted by our researchers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy

Exclusion Criteria:

* Pregnancy

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2013-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Body Weight | 3 1/2 year
  weight gain

CONTACTS AND LOCATIONS:
Locations (1):
- Dorms or student houseing, Ithaca, New York, United States